CLINICAL TRIAL: NCT04629222
Title: Tracheobronchitis May Constitute the Main Sign of Respiratory Involvement on the Lung SPECT/CT Images of COVID-19 Patients
Brief Title: Tracheobronchitis in Respiratory Involvement on the Lung SPECT/CT Images of Coronavirus Disease (COVID-19) Patients
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre Yves MARIE, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI154
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Infectious Disease of Lung
Keywords: Coronavirus Disease (COVID-19); Lung ventilation; Perfusion scintigraphy; Tracheobronchitis; Shortness of breath; Cadmium-Zinc-Telluride (CZT)-SPECT; Computer Tomography (CT)
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tracheobronchitis signs may be observed on ventilation lung scintigraphy during coronavirus disease (COVID-19) infection. This case report study aimed to analyze the rates and associated factors of such tracheobronchitis in COVID-19 patients referred to ventilation/perfusion lung scintigraphy with shortness of breath, suspected of pulmonary embolism.

DETAILED DESCRIPTION:
It was a retrospective study

ELIGIBILITY:
Inclusion Criteria:

* patient with Tracheobronchitis signs
* patient with lung scintigraphy exam

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients experiencing shortness of breath during the course of a COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Tracheobronchitis signs may be observed on ventilation lung scintigraphy during COVID-19 infection. | 1 month
  analyze the rates and associated factors of such tracheobronchitis in COVID-19 patients referred to ventilation/perfusion lung scintigraphy with shortness of breath, suspected of pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, France